CLINICAL TRIAL: NCT06176482
Title: Interventional Pilot Study on the Evaluation of the Functionality, the Safety, and the Reliability of an Implantable Bi-directional Myokinetic Interface for the Natural Control of Artificial Limbs
Brief Title: A Bidirectional MyoKinetic Implanted Interface for Natural Control of Artificial Limbs
Acronym: MYKY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Principal Investigator, Lorenzo Andreani, Clinical Professor, Azienda Ospedaliero, Universitaria Pisana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20084
Record Dates: First submitted 2023-11-08; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Upper Limb Amputation at the Wrist

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients enrolled and surgically treated (Experimental)
  Interventions: Device: Magnetic markers implantation

INTERVENTIONS:
Device: Magnetic markers implantation — Surgical implantation of magnetic markers in the upper limb stump to allow the management of an external hand prosthesis

SUMMARY:
This is a European project that it will develop an innovative robotic hand prosthesis, whose movements can be controlled in a natural and intuitive way. The project will be financed with 1.5 million euros by the European Research Council (ERC), through the "ERC Starting Grant 2015" program, one of the most competitive globally.

According to current approaches (even the most technologically advanced or still under development) the control of the movements of the prosthetic hand occurs on the decoding of the electrical potentials, transmitted by the brain and captured by the peripheral neuromuscular system, through electrodes. The project has the ambition of wanting to overcome the limits of these techniques, through the development of an interface based on magnetic markers implantable in the muscles, capable of monitoring the elongation (lengthening) of the residual muscles, as happens naturally when performing a task motor (action), for example grabbing a bottle. With this information MYKI wants to control the movements of a robotic hand in a natural and intuitive way. In terms of potential, magnetic markers could also be used to provide a sensory feedback to the person wearing the robotic prosthesis, when it interacts with the environment, just as happens in the natural hand.

DETAILED DESCRIPTION:
The 'MYKI- Studio Clinico' is a no-profit clinical study which aims at verifying the benefits and safety of an innovative upper limb interface, the Myokinetic interface, specifically conceived for patients with upper limb amputation. The study will verify whether the new interface, based on the use of implanted magnets, guarantees a natural and multi-degree of freedom control of robotic hands. Besides, the 'MYKI - Studio Clinico' will investigate if it is possible to convey physiologically appropriate proprioceptive information (i.e., movement and position information) of a missing finger or degrees of freedom through vibrations induced by implanted magnets. This idea is supported by the neuroscientific literature (Goodwin et al. 1972; Roll et al. 1989) and by studies conducted in the last years by the Sponsor's research group (see Clinical Investigator's Brochure ). Potential changes in the neurophysiological system will also be addressed. Finally, the controllability offered by the Myokinetic interface (i.e. the ability of the system to interpret the patient's voluntary motor commands, and to implement them on the robotic hand) will be experimentally compared with that offered by conventional surface electromyography (myoelectric prostheses).

The Myokinetic interface will produce a natural control and perception of robotic hands. The handbook "Manuale D'Uso" describes the instructions for the correct use of the device.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a uni- or bi-lateral trans-radial amputee.
* The patient had a traumatic amputation or a Congenital Hand Hypoplasia.
* The patient is 18 years or older, and younger than 70 years old.
* The amputation level guarantees to record muscle displacement and/or activity.
* The patient voluntarily accepts to receive the Myokinetic Interface.
* The patient voluntarily accepts to participate in all training and assessment sessions (follow-ups).

Exclusion Criteria:

* The patient is affected by peripheral vascular disease, neuropathies, or diabetes.
* The patient has current or prior dermatological conditions.
* The patient was diagnosed with a cognitive impairment, which prevents her/him from giving aware consent and following instructions.
* The patient has currently or had in the past psychological impairments (e.g., major personality disturbance, major depression, bipolar disorder).
* The patient has a history of or active substance abuse disorder.
* The patient has any concurrent disease or condition that might affect the treatment with the Myokinetic interface (e.g., neurological or musculoskeletal disorders).
* The patient is pregnant or lactating.
* The patient is participating in another study that can affect the outcome of this study.
* The patient is a wearer of an electronic device for the monitoring/treatment of vital functions (e.g., pacemaker or defibrillator), whose use might be affected by the electromagnetic field.
* The patient has to perform a magnetic resonance examination during the period of implantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pick and Lift Test (PLT) | Six weeks.
  The PLT measures motor coordination, i.e., the ability to coordinate the grip force and the load force while lifting an object, as well as the reliability of the recorded control signal while transporting the object. While the subject is sitting on a chair with the intact arm parallel to the trunk, and the amputated limb extending anteriorly on a table, he/she is asked to lift a small object from the table with the prosthesis.
Southampton Hand Assessment Procedure (SHAP) | Six weeks.
  The test consists of the sequential manipulation of 6 lightweight and 6 heavyweight abstract objects and 14 activities of daily living over a specific form-board. Lightweight objects should be manipulated first. The task involves pushing a button to start a timer, pick up and move the object from the rear slot to the front slot on the board, and complete the task by depressing the button on the timer again.
Minnesota Manual Dexterity Test (MMDT) | Six weeks.
  The objective of the test is to measure the capacity for simple but rapid eye-hand-finger movement as well as arm-hand movement and gross motor skills. It is a standardized test focused on coordination, which involves the use of a specific testing board that is placed on a table in front of the subject. There are holes in the board forming a rectangular grid, and the subject has to position some disks inside the holes according to a specific pattern of movements previously explained and demonstrated by the operator. A stopwatch is used in order to time the test.
Clothespin Relocation Test (CRT) | Six weeks.
  The objective is to evaluate the performance of a prosthetic user in a controlled environment and subsequently provide a measure of the expected functionality level of the user outside the laboratory/clinic. The user is instructed to allocate three clothespins between a horizontal rod and a vertical rod, and he/she is asked to fill out a post-test survey after five trials of the CRT.
Video recording in activities of the daily living (REC-ADL) | Six weeks.
  The objective is to evaluate the ability of the subject to carry out Activities of Daily Living (ADL) using the prosthesis. As an example, the subject can be instructed to hold a rubber ball in his/her hand and to maintain a stable grasp while moving the arm and shoulder in space.
Psychophysical test to understand the effect of vibration features on the elicited illusion of movement (VIB -FEATURES) | Six weeks.
  The objective of this study is to evaluate for each participant how vibration features (i.e., peak to peak amplitude, force, frequency, direction of the vibration) affect the participant perception and how we can improve the elicited illusion of movement in terms of vividness and range of motion. A psychophysical test will be conducted to determine the threshold of the parameters (frequency, amplitude, and vibration duration) in order to guarantee pleasant and effective sensory feedback.
Embodiment test - Rubber Hand Test (RHT) | Six weeks.
  The test evaluates for each participant how vibrations induced illusion of movement affect the embodiment (i.e., ownership and agency sensations) of a robotic hand when visual feedback, tactile feedback, and motor commands are congruently or incongruently delivered. Measurements of questionnaires and proprioceptive shift will be acquired to evaluate the embodiment.
Questionnaire for Phantom Limb (PLP) | Six weeks.
  The questionnaire evaluates the presence and the changes in PLP.
Ultrasound Imaging (US) | Six weeks.
  Evaluation of the contraction capability of residual muscles, the presence of fibrotic tissue, the presence of muscle atrophy.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ospedaliera Universitaria Pisana, Pisa, Pi, Italy

IPD SHARING:
Plan to Share IPD: No